CLINICAL TRIAL: NCT03316066
Title: Comparison of Two Volumes of Local Anesthetics on the Efficiency and Safety of Stellate Ganglion Block for the Treatment of Complex Regional Pain Syndrome of the Arm
Brief Title: Comparison of Volumes of Local Anesthetics on the Efficiency and Safety of Stellate Ganglion Block for CRPS of the Arm
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to recruit enough patients
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Veronique Brulotte, MD, MSc, FRCPC, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Maisonneuve RH
Record Dates: First submitted 2016-11-22; First posted 2017-10-20 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Complex Regional Pain Syndromes
Keywords: Stellate Ganglion; Local Anesthetic
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 5 (Experimental): stellate ganglion block with ropivacaine 0.2% 5 mL
  Interventions: Procedure: stellate ganglion block with ropivacaine 0.2% 5 mL
- Group 2 (Active Comparator): stellate ganglion block wit ropivacaine 0.2% 2 mL
  Interventions: Procedure: stellate ganglion block wit ropivacaine 0.2% 2 mL

INTERVENTIONS:
Procedure: stellate ganglion block with ropivacaine 0.2% 5 mL — Each patient will undergo two stellate ganglion blocks and receive both volumes of local anesthetics in random order. The stellate ganglion blocks will be separated by 3 weeks in order to assure that no residual effects from the previous block will influence the results.
  Arms: Group 5
Procedure: stellate ganglion block wit ropivacaine 0.2% 2 mL — Each patient will undergo two stellate ganglion blocks and receive both volumes of local anesthetics in random order. The stellate ganglion blocks will be separated by 3 weeks in order to assure that no residual effects from the previous block will influence the results.
  Arms: Group 2

SUMMARY:
The purpose of this study is to compare the efficiency and safety of 2ml versus 5ml of local anesthetics used in stellate ganglion blocks for the treatment of complex regional pain syndrome of the arm.

DETAILED DESCRIPTION:
To evaluate if 2ml of 0.2% ropivacaine is less effective in decreasing pain scores by more than 50% when compared to 5ml of 0.2% ropivacaine. To evaluate if 2ml of 0.2% ropivacaine is causes less side effects when compared to 5ml after a stellate ganglion block.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of complex regional pain syndrome of the arm according to the Budapest criteria and having already received a minimum of 3 stellate ganglion blocks. Only patients having received a minimum of 3 stellate ganglion blocks will be included since it is expected to have a progressive and sustained decrease in pain scores during the first 3 blocks.
* ASA 1 to 3 included

Exclusion Criteria:

* Patient refusal
* Contra-indications to the stellate ganglion block procedure such as coagulopathy, anticoagulants or anti platelet therapy other than aspirin, systemic or injection site infection, important neck deformity (post-radiotherapy or surgery, etc.), severe chronic obstructive pulmonary disease, contralateral diaphragm paralysis or contralateral pneumonectomy
* Allergy to local anesthetics
* Concomitant pain syndrome other than complex regional pain syndrome of the arm
* Liver or kidney failure (CrCl < 30 ml/min)
* Inability to understand à verbal numeric pain score scale after careful explanations
* Inability to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Pain score | 24 hours after the stellate ganglion block
  Evaluate the efficiency of stellate ganglion block in decreasing pain scores 24 hours after the procedure using a verbal numeric pain rating scale.

SECONDARY OUTCOMES:
Pain score | 7 days after the stellate ganglion block
  Evaluate the efficiency of stellate ganglion block in decreasing pain scores 7 days after the procedure using a verbal numeric pain rating scale.
Pain score | 14 days after the stellate ganglion block
  Evaluate the efficiency of stellate ganglion block in decreasing pain scores 14 days after the procedure using a verbal numeric pain rating scale.
Temperature increase in the ipsilateral arm | 1 hour after the procedure
  Evaluate the efficiency of stellate ganglion block on the increase in temperature of the ipsilateral arm using an infrared thermometer. The cutaneous temperature will be measured in order to determine the proportion of patients in each group reaching an increase of >1.5 C in the ipsilateral arm.
Horner Syndrome | 1 hour after the procedure
  Evaluate the efficiency of stellate ganglion block to produce an ipsilateral Horner Syndrome as defined by a ptosis and miosis. Evaluate the proportion of patients in each group presenting an ipsilateral Horner syndrome.
Occurrence of dysphagia after a stellate ganglion block | 1 hour after the procedure
  Patients describing having dysphagia after the stellate ganglion block
Occurrence of hoarseness after a stellate ganglion block | 1 hour after the procedure
  patients describing having hoarseness after a stellate ganglion block
Occurrence of foreign body sensation after a stellate ganglion block | 1h after the procedure
  patients describing having a foreign body sensation after the stellate ganglion block
Occurrence of dyspnea after a stellate ganglion block | 1h after the procedure
  patients describing having dyspnea after a stellate ganglion block
Occurrence of ipsilateral arm weakness after a stellate ganglion block | 1h after the procedure
  patients describing having ipsilateral arm weakness after a stellate ganglion block

OTHER OUTCOMES:
Occurrence of seizure during a stellate ganglion block | within 30 minutes of performing the stellate ganglion block
  patient having seizure
Occurrence of hematoma after a stellate ganglion block | During the first 7 days after the procedure
  physician or patient identifying a neck hematoma
Occurrence of pneumothorax after a stellate ganglion block | During the first 7 days after the procedure
  physician diagnosing a pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Brulotte, MD, Principal Investigator — Maisonneuve-Rosemont Hospital

IPD SHARING:
Plan to Share IPD: No